CLINICAL TRIAL: NCT01199679
Title: Evaluation of Distal Esophageal and Cardia Rubber Band Ligation and Mucosectomy in the Treatment of Subjects With Gastroesophageal Reflux Disease
Brief Title: Rubber Band Ligation and Mucosectomy for Gastroesophageal Reflux Disease (GERD)
Acronym: GERD
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 08-016
Record Dates: First submitted 2010-09-09; First posted 2010-09-13 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Gastroesophageal Reflux Disease; Heartburn; Regurgitation; Dyspepsia
Keywords: Gastroesophageal Reflux Disease; Heartburn; Regurgitation; Dyspepsia
MeSH Terms: conditions — Gastroesophageal Reflux; Heartburn; Dyspepsia

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Endoscopic Mucosal Resection (EMR) Group (Experimental)
  Interventions: Procedure: Mucosectomy
- Banding Group (Experimental)
  Interventions: Procedure: Rubber Band Ligation

INTERVENTIONS:
Procedure: Mucosectomy — Endoscopic mucosal resection in the upper GI tract.
  Arms: Endoscopic Mucosal Resection (EMR) Group
Procedure: Rubber Band Ligation — Endoscopically ligate esophageal varices at or above the gastroesophageal junction or to ligate internal hemorrhoids.
  Arms: Banding Group

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of two separate procedures to treat gastroesophageal reflux disease (GERD) also known as heartburn. The two therapies are: 1) a banding procedure alone using the Cook® 6 Shooter™ Saeed Multi-Band Ligator or 2) a banding/shaving procedure called Endoscopic Mucosal Resection (EMR) using the Cook® Duette™ Multi-Band Mucosectomy device.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older.
* Typical symptoms of heartburn and/or regurgitation requiring daily PPI therapy.
* Subject agrees to participate and signs consent form.

Exclusion Criteria:

* Patient is pregnant.
* Patient has a hiatal hernia greater than 2cm.
* Presence of persistent daily solid food dysphagia, unplanned weight loss over ten pounds, esophageal bleeding, or vomiting more than once per week).
* Active medical condition that would preclude the subject from finishing this study.
* BMI > 39.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2011-06; Primary Completion 2012-09 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Reduction of reflux symptoms measured by GERD HRQL | 6 months
  HRQL = Health Related Quality of Life Questionnaire

SECONDARY OUTCOMES:
Reduction in total esophageal acid exposure measured by 48 hour pH monitoring | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Glen A. Lehman, MD, Principal Investigator — Indiana University Hospital
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States